CLINICAL TRIAL: NCT06195150
Title: Overtaking Intra and Inter Tumoral Heterogeneity In Von Hippel-Lindau Related Renal Cancer
Acronym: ITHORinVHL
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Umberto Capitanio, Head of the Kidney Tumor Research Unit, IRCCS San Raffaele
Other Study IDs: PNRR-MR1-2022-12375818
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Clear Cell Renal Cell Carcinoma; VHL Syndrome
MeSH Terms: conditions — Carcinoma, Renal Cell; von Hippel-Lindau Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Pan-tumor histological assessment through molecular and histopathological evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VHL patients: Patients with hereditary Von Hippel-Lindau (VHL) with genetic diagnosis of VHL disease who have at least three tumors larger than 3cm that have to be surgically removed. The procedure involves standard surgery with the additional collection of 15ml of blood.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — 15ml of blood are harvested before surgery

SUMMARY:
The goal of this study is to comprehensively map intra and inter tumor heterogeneity of ccRCC in VHL patients through the use of imaging, molecular biology and genomics techniques.

DETAILED DESCRIPTION:
It was hypothesized that the high intra- inter-tumor heterogeneity of sporadic ccRCC also defines VHL-ccRCCs, including different lesions within individual patients, and it was assumed that decoding VHL-ccRCC heterogeneity by coupling imaging, histology and molecular profiling of multiregional biopsies would help improve diagnostic tests and therapeutic choices for VHL patients.

In order to comprehensively map intra and inter tumor heterogeneity of ccRCC in VHL patients, the aims of the study are:

1. To integrate pre-surgery imaging using conventional multiparametric MRI with tumor histology of geographical predeterminated multi-region biopsies in each ccRCC of VHL patients.
2. To combine multiplex immunohistochemistry, bulk and single cell RNA sequencing and somatic mutations analysis with pan-tumor histological assessment.
3. To optimize a protocol to generate VHL-ccRCC-derived tumor organoids (patient-derived organoids, PDO) and test anti tumor agents like HIF2alpha inhibitor in organoid cultures representative of intra- and inter-tumor heterogeneity.

This study will develop standardized models for diagnosis and molecular characterization of ccRCC in VHL disease using a combination of imaging, intrasurgical biopsying and multi-omics analysis. It will benefit of a clinical and research program devoted to VHL disease established at OSR in 2021 that centralizes Italian VHL patients. Since the current study relies on tumor biopsy techniques that are already established in clinical practice, the translational findings will be directly available and immediately affecting patients' care.

ELIGIBILITY:
Inclusion Criteria:

* VHL syndrome
* Presence of at least 3 kidney tumors larger that 3cm to be surgically removed

Exclusion Criteria:

* Absence of VHL
* Quantity of kidney tumors < 3
* Absence of surgery performance

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VHL patients with at least 3 kidney tumors larger that 3cm to be surgically removed
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Integrating Imaging and multiregion biopsy sampling in VHL related ccRCC | From month 3 to month 20
  Pre-surgery imaging will be integrated using conventional multiparametric MRI with tumor histology of geographical predeterminated multi-region biopsies in each ccRCC of VHL patients.
Determine immune and stromal heterogeneity in VHL-ccRCC | DNAseq and bulk RNAseq will be carried out from month 7 until month 20. Multiplex immunohistochemistry (IHC) in multiregional biopsies and standard IHC on the whole tumors will be performed the last 12 months of the study.
  Multiplex immunohistochemistry, bulk and single cell RNA sequencing and somatic mutations analysis with pan-tumor histological assessment will be combined.
Generation and characterization of VHL-ccRCC patient-derived organoids | From month 3 until the end of the project.
  A protocol to generate VHL-ccRCC-derived tumor organoids (patient-derived organoids, PDO) will be optimized to test anti tumor agents like HIF2alpha inhibitor in organoid cultures representative of intra- and inter-tumor heterogeneity.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy